CLINICAL TRIAL: NCT01629732
Title: Phase 2b Evaluation of PegIFNα Free Combinations of BMS-986094 (INX-08189) and Daclatasvir, With or Without Ribavirin, in Treatment Naive and Treatment Experienced Patients With Chronic Hepatitis C
Brief Title: Phase 2b Study of BMS-986094 and Daclatasvir, With or Without Ribavirin for the Treatment of Patients With Chronic Hepatitis C
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AI472-007; 2012-002519-24 (EudraCT Number)
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; BMS-986094; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Arm 1: Daclasasvir + BMS-986094 (100 mg) + Placebo (Experimental): Subjects will be re-randomized at Week 12 to complete therapy at this visit and enter post-treatment follow-up, or continue therapy for an additional 12 weeks (24 weeks of therapy)
  Re-Randomized Arm 1 to Arm 1a and 1b (additional 12 weeks treatment)
  Interventions: Drug: Daclatasvir; Drug: BMS-986094; Drug: Placebo for BMS-986094
- Arm 2: Daclasasvir + BMS-986094 (200 mg) (Experimental): Subjects will be re-randomized at Week 12 to complete therapy at this visit and enter post-treatment follow-up, or continue therapy for an additional 12 weeks (24 weeks of therapy)
  Re-Randomized Arm 2 to Arm 2a and 2b (additional 12 weeks treatment)
  Interventions: Drug: Daclatasvir; Drug: BMS-986094
- Arm 3: Daclasasvir + BMS-986094 (100 mg) + Placebo + Ribavirin (Experimental): Subjects will be re-randomized at Week 12 to complete therapy at this visit and enter post-treatment follow-up, or continue therapy for an additional 12 weeks (24 weeks of therapy)
  Re-Randomized Arm 3 to Arm 3a and 3b (additional 12 weeks treatment)
  Interventions: Drug: Daclatasvir; Drug: BMS-986094; Drug: Ribavirin; Drug: Placebo for BMS-986094
- Arm 4: Daclasasvir + BMS-986094 (200 mg) + Ribavirin (Experimental): Subjects will be re-randomized at Week 12 to complete therapy at this visit and enter post-treatment follow-up, or continue therapy for an additional 12 weeks (24 weeks of therapy)
  Re-Randomized Arm 4 to Arm 4a and 4b (additional 12 weeks treatment)
  Interventions: Drug: Daclatasvir; Drug: BMS-986094; Drug: Ribavirin
- Arm 5: Daclasasvir + BMS-986094 (200 mg) (Experimental): Genotype 1 PI-failure subjects
  Interventions: Drug: Daclatasvir; Drug: BMS-986094
- Arm 6: Daclasasvir + BMS-986094 (200 mg) (Experimental): Genotype 4 naive subjects
  Interventions: Drug: Daclatasvir; Drug: BMS-986094
- Arm 7: Daclasasvir + BMS-986094 (200 mg) (Experimental): Genotype 2/3 NR/relapse Subjects
  Interventions: Drug: Daclatasvir; Drug: BMS-986094

INTERVENTIONS:
Drug: Daclatasvir — Film coated tablet, Oral, 60 mg, Once daily, 12 or 24 weeks
  Other Names: BMS-790052 (DCV)
  Arms: Arm 1: Daclasasvir + BMS-986094 (100 mg) + Placebo; Arm 2: Daclasasvir + BMS-986094 (200 mg); Arm 3: Daclasasvir + BMS-986094 (100 mg) + Placebo + Ribavirin; Arm 4: Daclasasvir + BMS-986094 (200 mg) + Ribavirin
Drug: Daclatasvir — Film coated tablet, Oral, 60 mg, Once daily, 24 weeks
  Other Names: BMS-790052 (DCV)
  Arms: Arm 5: Daclasasvir + BMS-986094 (200 mg); Arm 6: Daclasasvir + BMS-986094 (200 mg); Arm 7: Daclasasvir + BMS-986094 (200 mg)
Drug: BMS-986094 — Capsule, Oral, 100 mg, Once daily, 12 or 24 weeks
  Arms: Arm 1: Daclasasvir + BMS-986094 (100 mg) + Placebo; Arm 3: Daclasasvir + BMS-986094 (100 mg) + Placebo + Ribavirin
Drug: BMS-986094 — Capsule, Oral, 200 mg, Once daily, 12 or 24 weeks
  Arms: Arm 2: Daclasasvir + BMS-986094 (200 mg); Arm 4: Daclasasvir + BMS-986094 (200 mg) + Ribavirin
Drug: BMS-986094 — Capsule, Oral, 200 mg, Once daily, 24 Weeks
  Arms: Arm 5: Daclasasvir + BMS-986094 (200 mg); Arm 6: Daclasasvir + BMS-986094 (200 mg); Arm 7: Daclasasvir + BMS-986094 (200 mg)
Drug: Ribavirin — Film coated tablet, Oral, 1000 mg or 1200 mg based on weight, Twice daily, 12 or 24 weeks
  Other Names: Copegus®
  Arms: Arm 3: Daclasasvir + BMS-986094 (100 mg) + Placebo + Ribavirin; Arm 4: Daclasasvir + BMS-986094 (200 mg) + Ribavirin
Drug: Placebo for BMS-986094 — Capsule, Oral, 0 mg, Once daily, 12 or 24 weeks
  Arms: Arm 1: Daclasasvir + BMS-986094 (100 mg) + Placebo; Arm 3: Daclasasvir + BMS-986094 (100 mg) + Placebo + Ribavirin

SUMMARY:
The purpose of this study is to evaluate the effectiveness of BMS-986094 and Daclatasvir (DCV) when given in combination with or without Ribavirin

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ≥ 18 years of age
* Subjects chronically infected with Hepatitis C virus (HCV) genotype 1,2,3 or 4
* HCV RNA viral load ≥ 10,000 IU/mL
* Subjects with compensated cirrhosis are permitted (compensated cirrhotics are capped at approximately 25% of treated population)
* Body Mass Index (BMI) of 18 to 35 kg/m2
* Seronegative for Hepatitis C virus (HIV) and Hepatitis B

Exclusion Criteria:

* Evidence of decompensated liver disease
* Evidence of medical condition contributing to chronic liver disease other than HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2014-02 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with SVR4 defined as HCV RNA < LOQ (25 IU/mL; detectable or undetectable) at 4 weeks post treatment to be evaluated in GT1 (naive and NR) subjects randomized to the 12-week treatment arm (arms 1a, 2a, 3a, 4a) | Follow up Week 4
  * SVR = Sustained virologic response
  * HCV = Hepatitis C virus
  * RNA = Ribonucleic acid
  * LOQ = Limit of quantitation

SECONDARY OUTCOMES:
Proportion of treated subjects with SVR4 in genotype (GT) 1 naive and non-responder (NR) subjects randomized to the 24-week treatment arms (arms 1b, 2b, 3b, 4b) | Follow up Week 4 (SVR4)
Proportion of treated subjects with SVR4 in genotype 1 protease inhibitor (PI)failures, genotype 4 naive, and genotype 2/3 NR/relapse subjects (arms 5, 6, 7) | Follow up Week 4 (SVR4)
Proportion of treated subjects in each study population (GT1 naive, GT1 NR, or GT1 PI-failure, GT4 naive, GT2/3 NR/relapse), for each regimen and duration, who achieve HCV RNA < LOQ at post-treatment | Post-treatment Week 2 (SVR2), Week 8 (SVR8), Week 12 (SVR12), Week 24 (SVR24), and Week 36 (SVR36, for the 12 week arms)
Proportion of treated subjects in each study population, by regimen, who achieve HCV RNA < LOQ (detectable/undetectable) | Weeks 1, 2, 4, 6, 8, 12 and End of Treatment (Week 12 or 24)
Proportion of subjects in each study population, be regimen, who achieve HCV RNA undetectable | Weeks 1, 2, 4, 6, 8, 12 and End of Treatment (Week 12 or 24)
Safety and tolerability of BMS-986094 and DCV ± RBV as measured by the frequency of deaths, serious adverse events (SAEs), discontinuations due to Adverse Events (AEs), and severity Grade 3/4 laboratory abnormalities | Up to post treatment Week 36

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Orlando, Florida, United States

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx